CLINICAL TRIAL: NCT03182244
Title: Phase 3 Open-label, Multicenter, Randomized Study of ASP2215 Versus Salvage Chemotherapy in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML) With FLT3 Mutation
Brief Title: A Study of ASP2215 Versus Salvage Chemotherapy In Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML) With FMS-like Tyrosine Kinase 3 (FLT3) Mutation
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2215-CL-0303; CTR20170326 (Registry Identifier: Chinadrugtrials.org.cn)
Record Dates: First submitted 2017-06-08; First posted 2017-06-09 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: AML With FLT3 Mutation
Keywords: gilteritinib; Acute Myeloid Leukemia (AML); ASP2215
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib; Cytarabine; Mitoxantrone; Etoposide; Granulocyte Colony-Stimulating Factor; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gilteritinib (Experimental): Participants received 120 milligrams (mg) gilteritinib (3 tablets of 40 mg) orally, once a day in continuous 28-day cycles until treatment discontinuation criteria were met. Participants who met the treatment discontinuation criteria, entered the long-term follow-up period. Participants remained in the long-term follow-up period for up to 3 years from the participant's end of treatment visit or until discontinuation from the study.
  Interventions: Drug: Gilteritinib
- Salvage chemotherapy (Active Comparator): Participants received salvage chemotherapy in continuous 28-day cycles per institutional guidelines:LoDAC:20mg cytarabine twice daily SC/IV for 10 days. MEC:mitoxantrone 6 milligrams per square meter(mg/m^2)/day IV for 5 days (days 1 to 5), etoposide 100mg/m^2/day IV for 5 days (days 1 to 5), cytarabine 1000mg/m^2/day IV for 5 days (days 1 to 5). FLAG: granulocyte colony-stimulating factor (G-CSF) 300 micrograms per square meter (μg/m^2) per day SC/IV for 5 days (days 1 to 5), fludarabine 30mg/m^2/day IV for 5 days (days 2 to 6), cytarabine 2000mg/m^2/day IV for 5 days (days 2 to 6). Participants meeting treatment discontinuation criteria, entered long-term follow-up, for up to 3 years from end of treatment visit/until study discontinuation. Based on interim analysis outcome, at investigators discretion, treatment period participants had option to enter crossover extension to receive 120mg gilteritinib, orally, once daily in continuous 28-day cycles until treatment discontinuation.
  Interventions: Drug: Cytarabine; Drug: Mitoxantrone; Drug: Etoposide; Drug: G-CSF; Drug: Fludarabine

INTERVENTIONS:
Drug: Gilteritinib — Tablet administered orally once daily.
  Other Names: ASP2215
  Arms: Gilteritinib
Drug: Cytarabine — Once/twice daily Intravenously (IV)/subcutaneously (SC).
  Arms: Salvage chemotherapy
Drug: Mitoxantrone — Once daily IV injection.
  Arms: Salvage chemotherapy
Drug: Etoposide — Once daily IV injection.
  Arms: Salvage chemotherapy
Drug: G-CSF — Once daily IV/SC injection.
  Arms: Salvage chemotherapy
Drug: Fludarabine — Once daily IV injection.
  Arms: Salvage chemotherapy

SUMMARY:
The purpose of this study was to determine the clinical benefit of ASP2215 therapy in participants with FMS-like tyrosine kinase (FLT3) mutated AML who were refractory to or had relapse after first-line AML therapy as shown with overall survival (OS) compared to salvage chemotherapy. In addition, this study evaluated safety as well as determined the overall efficacy in event-free survival (EFS) and complete remission (CR) rate of ASP2215 compared to salvage chemotherapy.

DETAILED DESCRIPTION:
Participants considered an adult according to local regulations at the time of signing informed consent were randomized in a 1:1 ratio and received ASP2215 or salvage chemotherapy. Participants entered the screening period up to 14 days prior to the start of treatment. Prior to randomization, the investigator preselected a salvage chemotherapy regimen for each participant; options included low-dose cytarabine (LoDAC), mitoxantrone, etoposide and intermediate-dose cytarabine (MEC) or fludarabine, high-dose cytarabine and granulocyte colony-stimulating factor (FLAG). The randomization was stratified by response to first-line therapy and preselected salvage chemotherapy. Participants were administered treatment over continuous 28-day cycles.

Among the participants, approximately 20 Chinese participants who were randomized into the ASP2215 arm were allocated to the pharmacokinetic (PK) cohort. Participants in the PK cohort were requested to be hospitalized from the date of randomization (Day 1) to at least the completion of all the assessments planned on Day 2. All participants in the PK cohort underwent blood sampling for PK measurement of ASP2215. Participants in PK cohort were administered the study drug in the same manner and underwent the same efficacy and safety assessments as other participants except for blood sampling for additional PK measurements.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of primary AML or AML secondary to myelodysplastic syndrome (MDS) according to World Health Organization (WHO) classification as determined by pathology review at the treating institution.
* Participant is refractory to or relapsed after first-line AML therapy (with or without HSCT)

  * Refractory to first-line AML therapy is defined as:

    a. Participant did not achieve CR/CRi/CRp under initial therapy. A participant eligible for standard therapy must receive at least 1 cycle of an anthracycline containing induction block in standard dose for the selected induction regimen. A participant not eligible for standard therapy must have received at least 1 complete block of induction therapy seen as the optimum choice of therapy to induce remission for this participant.
  * Untreated first hematologic relapse is defined as:

    1. Participant must have achieved a CR/CRi/CRp with first-line treatment and has hematologic relapse.
* Participant is positive for FLT3 mutation in bone marrow or whole blood as determined by the central lab. A participant with rapidly proliferative disease and unable to wait for the central lab results can be enrolled based on a local test performed after completion of the last interventional treatment. Participants can be enrolled from a local test result if the participants have any of the following FLT3 mutations: FLT3-internal tandem duplication (ITD), FLT3-tyrosine kinase domain (TKD)/D835 or FLT3-TKD/I836.
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Participant is eligible for preselected salvage chemotherapy.
* Participant must meet the following criteria as indicated on the clinical laboratory tests:

  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN)
  * Serum total bilirubin (TBL) ≤ 1.5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or an estimated glomerular filtration rate of > 50 mL/min as calculated by the Modification of Diet in Renal Disease equation.
* Participant is suitable for oral administration of study drug.
* Participant agrees not to participate in another interventional study while on treatment.

Inclusion Criteria for COE:

Participant is eligible for the COE if they continue to meet all inclusion criteria from the main protocol in addition to the following when the participant is evaluated for eligibility to participate in the COE portion of the study:

* Participant has received study treatment of either LoDAC, MEC or FLAG and has no response or progressive disease.
* Participant have not received other antileukemic therapy after EOT (hydroxyurea is allowed for the control of peripheral leukemic blasts in participants with leukocytosis).
* Participant agrees not to participate in another interventional study while on treatment.

Exclusion Criteria:

* Participant was diagnosed as acute promyelocytic leukemia.
* Participant has BCR-ABL-positive leukemia (chronic myelogenous leukemia in blast crisis).
* Participant has AML secondary to prior chemotherapy for other neoplasms (except for MDS).
* Participant is in second or later hematologic relapse or has received salvage therapy for refractory disease.
* Participant has clinically active central nervous system leukemia..
* Participant has been diagnosed with another malignancy, unless disease-free for at least 5 years. Participants with treated nonmelanoma skin cancer, in situ carcinoma or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed. Participants with organ-confined prostate cancer with no evidence of recurrent or progressive disease are eligible if hormonal therapy has been initiated or the malignancy has been surgically removed or treated with definitive radiotherapy.
* Participant has received prior treatment with ASP2215 or other FLT3 inhibitors (with the exception of sorafenib and midostaurin used in first-line therapy regimen as part of induction, consolidation and/or maintenance).
* Participant has clinically significant abnormality of coagulation profile, such as disseminated intravascular coagulation.
* Participant has had major surgery within 4 weeks prior to the first study dose.
* Participant has radiation therapy within 4 weeks prior to the first study dose.
* Participant has congestive heart failure New York Heart Association (NYHA) class 3 or 4 or participant with a history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram (ECHO) performed within 1 month prior to study entry results in a left ventricular ejection fraction (LVEF) that is ≥ 45%.
* Participant with mean of triplicate Fridericia-corrected QT interval (QTcF) > 450 ms at Screening based on central reading.
* Participant with Long QT Syndrome at Screening.
* Participant with hypokalemia and hypomagnesemia at Screening (defined as values below lower limit of normal [LLN]).
* Participant requires treatment with concomitant drugs that are strong inducers of CYP3A.
* Participant requires treatment with concomitant drugs that are strong inhibitors or inducers of P-gp with the exception of drugs that are considered absolutely essential for the care of the participant.
* Participant requires treatment with concomitant drugs that target serotonin 5-hydroxytryptamine receptor 1 (5HT1R) or 5-hydroxytryptamine receptor 2B (5HT2BR) receptors or sigma nonspecific receptor with the exception of drugs that are considered absolutely essential for the care of the participant.
* Participant has an active uncontrolled infection.
* Participant is known to have human immunodeficiency virus infection.
* Participant has active hepatitis B or C or other active hepatic disorder.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has active clinically significant (graft-versus-host disease) GVHD or is on treatment with systemic corticosteroids for GVHD.
* Participant has an FLT3 mutation other than the following: FLT3-ITD, FLT3-TKD/D835 or FLT3-TKD/I836.

Exclusion Criteria for COE:

Participant will be excluded from participation in the COE if they meet any of the exclusion criteria listed in the main protocol or when the participant is evaluated for eligibility to participate in the COE portion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (49):
- China (28):
  - Site CN103, Beijing
  - Site CN108, Beijing
  - Site CN109, Beijing
  - Site CN110, Beijing
  - Site CN131, Beijing
  - Site CN116, Changchun
  - Site CN120, Changsha
  - Site CN119, Fuzhou
  - Site CN102, Guangzhou
  - Site CN114, Guangzhou
  - Site CN121, Guangzhou
  - Site CN130, Guiyang
  - Site CN107, Hangzhou
  - Site CN118, Hefei
  - Site CN123, Huangpu Qu
  - Site CN117, Jinan
  - Site CN133, Lanzhou
  - Site CN128, Nanjing
  - Site CN106, Qingdao
  - Site CN126, Shanghai
  - Site CN129, Shanghai
  - Site CN125, Shenyang
  - Site CN101, Tianjin
  - Site CN105, Wuhan
  - Site CN122, Xi'an
  - Site CN132, Zhangzhou
  - Site CN113, Zhengzhou
  - Site CN136, Zhengzhou
- Malaysia (6):
  - Site MY306, Ampang
  - Site MY305, George Town
  - Site MY301, Johor Bahru
  - Site MY304, Kota Kinabalu
  - Site MY302, Kuala Lumpur
  - Site MY303, Pulau Pinang
- Russia (7):
  - Site RU506, Kemerovo
  - Site RU504, Krasnoyarsk
  - Site RU508, Moscow
  - Site RU509, Moscow
  - Site RU501, Saint Petersburg
  - Site RU502, Saint Petersburg
  - Site RU507, Saint Petersburg
- Singapore (3):
  - Site SG401, Singapore
  - Site SG402, Singapore
  - Site SG403, Singapore
- Thailand (5):
  - Site TH203, Bangkok
  - Site TH205, Bangkok
  - Site TH204, Chiang Mai
  - Site TH201, Khon Kaen
  - Site TH202, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Jiang B, Li J, Liu L, Du X, Jiang H, Hu J, Zeng X, Sakatani T, Kosako M, Deng Y, Girshova L, Bondarenko S, Lee LWL, Khuhapinant A, Martynova E, Hasabou N, Wang J. Gilteritinib versus salvage chemotherapy in predominantly Asian patients with relapsed/refractory FLT3-mutated acute myeloid leukemia: a regional analysis of COMMODORE in China, South-East Asia, and Russia. Ann Hematol. 2025 Mar;104(3):1563-1575. doi: 10.1007/s00277-025-06235-y. Epub 2025 Mar 10. PMID 40063243

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with FMS-like tyrosine kinase 3 (FLT3) mutations with relapsed or refractory Acute Myeloid Leukemia (AML) after first-line therapy were enrolled for this study.
  21 participants from six china sites were included in Giltertinib PK cohort.
Pre-assignment Details: Randomization was stratified by response to first-line therapy and preselected salvage chemotherapy.
  Results were reported up to primary analysis data cut-off of 25 December 2023 (approximately 74 months).
Groups:
- Salvage Chemotherapy: Participants received salvage chemotherapy in continuous 28-day cycles per institutional guidelines.
  Salvage chemotherapy included:
  Low dose cytarabine (LoDAC): 20 mg cytarabine administered twice daily by subcutaneous (SC)/intravenous (IV) injection for 10 days.
  Mitoxantrone, etoposide and intermediate dose cytarabine (MEC): mitoxantrone 6 milligrams per square meter(mg/m^2) per day administered by IV for 5 days (days 1 through 5), etoposide 100 mg/m^2 per day administered by IV for 5 days (days 1 through 5), cytarabine 1000 mg/m^2 per day administered by IV for 5 days (days 1 through 5).
  Fludarabine, cytarabine and granulocyte colony-stimulating factor (FLAG): granulocyte colony-stimulating factor (G-CSF) 300 micrograms per square meter (μg/m^2) per day administered by SC/IV for 5 days (days 1 through 5), fludarabine 30 mg/m^2 per day administered by IV for 5 days (days 2 through 6), cytarabine 2000 mg/m^2 per day administered by IV for 5 days (days 2 through 6). Participants who met treatment discontinuation criteria, entered long-term follow-up and remained in the period for up to 3 years from the participant's end of treatment visit/until discontinuation from study.
  Based on the outcome of interim analysis, at investigators discretion, participants in the treatment period had the option to enter crossover extension (COE) period to receive 120 mg gilteritinib, orally, once a day in continuous 28-day cycles until treatment discontinuation criteria was met.
Period: Treatment Period (Upto 1917 Days)
Arm/Group | Gilteritinib | Salvage Chemotherapy
Started | 137 | 139
LoDAC | 0 | 27
MEC | 0 | 42
FLAG | 0 | 70
Chinese PK Cohort | 21 | 0
Completed | 0 | 26
Not Completed | 137 | 113
Not completed — Adverse Event | 8 | 9
Not completed — Death | 19 | 8
Not completed — Miscellaneous | 12 | 0
Not completed — Disease Relapse | 41 | 5
Not completed — Physician Decision | 5 | 10
Not completed — Withdrawal by Subject | 10 | 28
Not completed — Protocol Violation | 4 | 1
Not completed — Progressive Disease | 18 | 9
Not completed — Lack of Efficacy | 20 | 43
Period: Long Term Follow-up (Up to 1232 Days)
Arm/Group | Gilteritinib | Salvage Chemotherapy
Started | 100 (37 participants did not enter the long term follow up period for this arm.) | 105 (34 participants did not enter the long term follow up period for this arm.)
Completed | 9 | 12
Not Completed | 91 | 93
Not completed — Miscellaneous | 4 | 3
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Lost to Follow-up | 6 | 7
Not completed — Death | 76 | 75
Period: Cross Over Extension (COE) Period
Arm/Group | Gilteritinib | Salvage Chemotherapy
Started | 0 (None of the participants from Salvage chemotherapy entered the COE period.) | 0 (None of the participants from Salvage chemotherapy entered the COE period.)
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat analysis Set (ITT) : The ITT consisted of all participants who were randomized.
Groups:
- Gilteritinib: Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day in continuous 28-day cycles until treatment discontinuation criteria were met. Participants who met the treatment discontinuation criteria, entered the long-term follow-up period. Participants remained in the long-term follow-up period for up to 3 years from the participant's end of treatment visit or until discontinuation from the study.
- Salvage Chemotherapy: Participants received salvage chemotherapy in continuous 28-day cycles per institutional guidelines.
  Salvage chemotherapy included:
  LoDAC: 20 mg cytarabine administered twice daily by SC/IV injection for 10 days.
  MEC: mitoxantrone 6 mg/m^2 per day administered by IV for 5 days (days 1 through 5), etoposide 100 mg/m^2 per day administered by IV for 5 days (days 1 through 5), cytarabine 1000 mg/m^2 per day administered by IV for 5 days (days 1 through 5).
  FLAG: G-CSF 300 μg/m^2 per day administered by SC/IV for 5 days (days 1 through 5), fludarabine 30 mg/m^2 per day administered by IV for 5 days (days 2 through 6), cytarabine 2000 mg/m^2 per day administered by IV for 5 days (days 2 through 6). Participants who met treatment discontinuation criteria, entered long-term follow-up and remained in the period for up to 3 years from the participant's end of treatment visit/until discontinuation from study.
  Based on the outcome of interim analysis, at investigators discretion, participants in the treatment period had the option to enter COE period to receive 120 mg gilteritinib, orally, once a day in continuous 28-day cycles until treatment discontinuation criteria was met.
- Total: Total of all reporting groups
Arm/Group | Gilteritinib | Salvage Chemotherapy | Total
Number analyzed (Participants) | 137 | 139 | 276
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.9 (16.2) | 46.2 (15.1) | 46.6 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 70 | 146
  Male | 61 | 69 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 136 | 139 | 275
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 123 | 120 | 243
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 19 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 90 | 92 | 182
  Russia | 14 | 19 | 33
  Malaysia | 15 | 14 | 29
  Thailand | 14 | 10 | 24
  Singapore | 4 | 4 | 8
Response to First-Line Therapy [Number; unit: Participants]
  Relapse within 6 months after allogeneic HSCT | 1 | 4 | 5
  Relapse after 6 months after allogeneic HSCT | 2 | 2 | 4
  Primary refractory without HSCT | 80 | 81 | 161
  Relapse within 6 months after CRc and no HSCT | 31 | 29 | 60
  Relapse after 6 months after CRc and no HSCT | 23 | 23 | 46
Preselected Salvage Chemotherapy [Number; unit: Participants]
  High intensity chemotherapy | 110 | 112 | 222
  Low intensity chemotherapy | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death due to any cause. Participants who were still alive or lost to follow up were censored at the time they were last known to be alive. Kaplan-Meier (KM) estimates was used for analysis.
Time Frame: From the date of randomization up to the date of death (up to approximatley 74 months)
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 137 | 139
months | 10.3 [8.8 to 12.7] | 5.4 [4.1 to 8.1]
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Test type: Superiority; p = 0.00152, Log Rank; Stratification factors were response to first-line AML therapy and preselected salvage chemotherapy per interactive response technology (IRT); Hazard Ratio (HR) = 0.612, 95% CI 2-sided [0.451 to 0.832] — Based on Cox proportional hazard model. Assuming proportional hazards, an HR < 1 indicates a reduction in hazard rate where the numerator is the Gilteritinib arm and the denominator is the Salvage chemotherapy arm

2. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS: time from the date of randomization until the date of documented relapse, treatment failure, death, reported off treatment relapse or new AML therapy start whichever occued first, including the long-term follow-up data. KM estimate was used for analysis.
  Relapse was defined as documentation of any of following events:
  * Bone marrow (BM) blasts ≥ 5% (not attributable to regenerating BM)
  * Reappearance or new appearance of extramedullary leukemia
  * Reappearance of significant numbers of peripheral blasts
  Treatment failure: Treatment failure was defined as participant who ends treatment without having a previous response of CR, CR with incomplete platelet recovery (CRp) and CR with incomplete hematological recover (CRi).
Time Frame: From the date of randomization up to the date of documented relapse, treatment failure or death from any cause, off-treatment relapse and start of new AML therapy (up to approximately 74 months)
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 137 | 139
months | 2.1 [0.1 to 3.2] | 0.6 [0.2 to 1.2]
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Test type: Superiority; p = 0.00005, Log Rank; Stratification factors were response to first-line AML therapy and preselected salvage chemotherapy per IRT; Hazard Ratio (HR) = 0.589, 95% CI 2-sided [0.438 to 0.792] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Complete Remission (CR) Rate
Description: Percentage of participants with CR were reported. CR: morphologically leukemia-free state, with absolute neutrophil count (ANC) > 1x10^9 per liter (1x10^9/L), platelet count ≥ 100x10^9/L and normal marrow differential with <5% blasts. They were red blood cell (RBC) and platelet transfusion independent and no evidence of extramedullary leukemia or Auer rods was necessary.
Time Frame: From the date of randomization up to approximately 74 months
Population: ITT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 137 | 139
Percentage of participants | 20.4 [14.0 to 28.2] | 11.5 [6.7 to 18.0]
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Test type: Superiority; p = 0.04256, Cochran-Mantel-Haenszel; Stratification factors: first-line AML therapy & preselected salvage chemotherapy/IRT response. Treatment difference based on stratification factors; Treatment difference = 8.9, 95% CI 2-sided [0.3 to 17.5]

4. Secondary Outcome: Duration of CR
Description: Duration of CR: time from the date of achieving first CR until date of first documented relapse for participants who achieved CR. KM estimate was used for analysis.
  CR: morphologically leukemia-free state, with ANC> 1x10^9/L, platelet count ≥ 100x10^9/L and normal marrow differential with < 5% blasts. They were RBC and platelet transfusion independent and no evidence of extramedullary leukemia.
  Relapse was defined as documentation of any of following events:
  * BM blasts ≥ 5% (not attributable to regenerating BM)
  * Reappearance or new appearance of extramedullary leukemia
  * Reappearance of significant numbers of peripheral blasts
Time Frame: From date of achieving CR until date of confirmed relapse (maximum duration was 53.4 months )
Population: ITT. Participants with CR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 28 | 16
months | 24.0 [4.6 to NA] — Upper limit of confidence interval was not estimable due to an insufficient number of events to determine 50% survival. | NA [1.0 to NA] — Median and upper limit of confidence interval was not estimable due to an insufficient number of events to determine 50% survival.
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Test type: Superiority; p = 0.88710, Log Rank; Stratification factors were response to first-line AML therapy and preselected salvage chemotherapy per IRT; Hazard Ratio (HR) = 1.163, 95% CI 2-sided [0.131 to 10.338] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Duration of Composite Complete Remission (CRc)
Description: Duration of CRc: time from date of achieving first CRc until date of first documented relapse for participants who achieved CRc. KM estimate was used for analysis.
  CRc: rate of all complete & incomplete remissions [CR + CRp + CRi]. CR: morphologically leukemia-free state, with ANC> 1x10^9/L, platelet count ≥ 100x10^9/L and normal marrow differential with <5% blasts. They were RBC and platelet transfusion independent and no evidence of extramedullary leukemia.
  CRp: met all CR criteria except incomplete platelet recovery (< 100x10^9/L). CRi: met all CR criteria, except for incomplete hematological recovery with residual neutropenia < 1x10^9/L with or without complete platelet recovery.
  Relapse: BM blasts ≥ 5%, reappearance or new appearance of extramedullary leukemia, reappearance of significant numbers of peripheral blasts.
Time Frame: From date of achieving CRc until date of confirmed relapse (maximum duration was 60 months)
Population: ITT. Participants with best overall response of CRc were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 73 | 31
months | 4.1 [2.8 to 5.6] | NA [NA to NA] — Median, upper and lower limit of confidence interval were not estimable due to an insufficient number of events to determine 50% survival.
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Test type: Superiority; p = 0.55969, Log Rank; Stratification factors were response to first-line AML therapy and preselected salvage chemotherapy per IRT; Hazard Ratio (HR) = 0.710, 95% CI 2-sided [0.209 to 2.414] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Duration of CR/Complete Remission With Partial Hematologic Recovery (CRh)
Description: Duration of CR/CRh: time from date of achieving first CR/CRh until date of first documented relapse for participants who achieved CR/CRh. KM estimate was used for analysis.
  CR: morphologically leukemia-free state, with ANC> 1x10^9/L, platelet count ≥ 100x10^9/L and normal marrow differential with <5% blasts. They were RBC and platelet transfusion independent and no evidence of extramedullary leukemia.
  CRh was defined as a condition at the post baseline visit, having bone marrow blasts < 5%, partial hematologic recovery ANC ≥ 0.5x10^9/L and platelets ≥ 50x10^9/L, no evidence of extramedullary leukemia and cannot be classified as CR. The blast counts in peripheral blood was ≤ 2%.
  Relapse: BM blasts ≥ 5%, reappearance or new appearance of extramedullary leukemia, reappearance of significant numbers of peripheral blasts.
Time Frame: From date of achieving CR/CRh until date of confirmed relapse (maximum duration was 58.1 months)
Population: ITT. Participants with CR/CRh were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 44 | 20
months | 5.6 [2.8 to 24.0] | NA [NA to NA] — Upper and lower limits of confidence interval was not estimable due to an insufficient number of events to determine 50% survival.
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Test type: Superiority; p = 0.66261, Log Rank; Stratification factors were response to first-line AML therapy and preselected salvage chemotherapy per IRT; Hazard Ratio (HR) = 1.583, 95% CI 2-sided [0.192 to 13.048] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Duration Of Response (DOR)
Description: DOR: time from date of first CRc (CR+CRp+CRi)/PR until date of first documented relapse for participants who achieved CRc or PR. KM estimate used for analysis.
  CR: morphologically leukemia-free state, with ANC> 1x10^9/L, platelet count ≥ 100x10^9/L and normal marrow differential with <5% blasts. They were RBC and platelet transfusion independent and no evidence of extramedullary leukemia.
  CRp: met all CR criteria except incomplete platelet recovery (< 100x10^9/L). CRi: met all CR criteria, except for incomplete hematological recovery with residual neutropenia < 1x10^9/L with or without complete platelet recovery.
  PR: condition with regeneration of normal hematopoietic cells in BM, no detectable blasts, ≥ 50% decrease of blasts in BM aspirate & total BM blasts of 5-25%.
  Relapse: BM blasts ≥ 5%, reappearance or new appearance of extramedullary leukemia, reappearance of significant numbers of peripheral blasts and increase in the percentage of blasts in the BM aspirate to > 25%.
Time Frame: From date of achieving CRc/PR until date of confirmed relapse (maximum duration was 52.1 months)
Population: ITT. Participants with best overall response of CRc/PR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 93 | 38
months | 3.7 [2.5 to 4.7] | NA [1.2 to NA] — Median and lower limit of confidence interval was not estimable due to an insufficient number of events to determine 50% survival.
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Test type: Superiority; p = 0.55731, Log Rank; Stratification factors were response to first-line AML therapy and preselected salvage chemotherapy per IRT; Hazard Ratio (HR) = 0.756, 95% CI 2-sided [0.286 to 1.999] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: CR/CRh Rate
Description: Percentage of participants with CR/CRh was reported. CR: morphologically leukemia-free state, with ANC> 1x10^9/L, platelet count ≥ 100x10^9/L and normal marrow differential with <5% blasts. They were RBC and platelet transfusion independent and no evidence of extramedullary leukemia.
  CRh was defined as a condition at the post baseline visit, having bone marrow blasts < 5%, partial hematologic recovery ANC ≥ 0.5x10^9/L and platelets ≥ 50x10^9/L, no evidence of extramedullary leukemia and could be classified as CR. The blast counts in peripheral blood was ≤ 2%.
Time Frame: From the date of randomization up to approximately 74 months
Population: ITT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 137 | 139
Percentage of participants | 32.1 [24.4 to 40.6] | 14.4 [9.0 to 21.3]
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Test type: Superiority; p = 0.00049, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Treatment difference = 17.7, 95% CI 2-sided [7.9 to 27.5]

9. Secondary Outcome: Best Response Rate
Description: Defined as percentage of participants with CR, CRp, CRi, PR, no response (NR) & not estimable (NE). CR: morphologically leukemia-free state, with ANC> 1x10^9/L, platelet count ≥ 100x10^9/L & normal marrow differential with < 5% blasts. They were RBC & platelet transfusion independent & no evidence of extramedullary leukemia. CRp: met all CR criteria except incomplete platelet recovery (<100x10^9/L). CRi: met all CR criteria, except incomplete hematological recovery with residual neutropenia < 1x10^9/L with/without complete platelet recovery. PR: condition with regeneration of normal hematopoietic cells in BM, no detectable blasts, ≥ 50% decrease of blasts in BM aspirate & total BM blasts of 5-25%. <=5% BM blasts if Auer rods are present, no evidence of extramedullary leukemia. Not Estimable (NE): No BM assessed/no myeloblast value, no blast value from peripheral blood or ≤2%, & no extramedullary leukemia. No Response (NR): Response not categorized as CR, CRp, CRi, PR or NE.
Time Frame: From the date of randomization up to approximately 74 months
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 137 | 139
Percentage of participants
  CR | 20.4 | 11.5
  CRp | 13.1 | 0.7
  CRi | 19.7 | 10.1
  PR | 14.6 | 5.0
  NR | 27.7 | 34.5
  NE | 4.4 | 38.1

10. Secondary Outcome: Leukemia-Fee Survival (LFS)
Description: LFS: time from the date of first CRc (CR+CRp+CRi) until the date of documented relapse or death for participants who achieved CRc.
  CR: morphologically leukemia-free state, with ANC> 1x10^9/L, platelet count ≥ 100x10^9/L and normal marrow differential with < 5% blasts. They were RBC and platelet transfusion independent and no evidence of extramedullary leukemia.
  CRp: met all CR criteria except incomplete platelet recovery (< 100x10^9/L). CRi: met all CR criteria, except for incomplete hematological recovery with residual neutropenia < 1x10^9/L with or without complete platelet recovery.
  Relapse: BM blasts ≥ 5%, reappearance or new appearance of extramedullary leukemia, reappearance of significant numbers of peripheral blasts.
Time Frame: From first day of achieving first CRc to the first day of confirmed relapse/death (maximum duration was 60.0 months)
Population: ITT. Participants with best overall response of CRc were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 73 | 31
months | 3.9 [2.8 to 5.4] | 6.9 [2.9 to 10.4]
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Test type: Superiority; p = 0.56944, Log Rank; Stratification factors were response to first-line AML therapy and preselected salvage chemotherapy per IRT; Hazard Ratio (HR) = 0.857, 95% CI 2-sided [0.494 to 1.487] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Composite Complete Remission (CRc)
Description: Percentage of participants with CRc (CR+CRp+CRi) was reported. CR: morphologically leukemia-free state, with ANC> 1x10^9/L, platelet count ≥ 100x10^9/L and normal marrow differential with <5% blasts. They were RBC and platelet transfusion independent and no evidence of extramedullary leukemia.
  CRp: met all CR criteria except incomplete platelet recovery (< 100x10^9/L). CRi: met all CR criteria, except for incomplete hematological recovery with residual neutropenia < 1x10^9/L with or without complete platelet recovery.
Time Frame: From the date of randomization up to approximately 74 months
Population: ITT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Salvage Chemotherapy: PParticipants received salvage chemotherapy in continuous 28-day cycles per institutional guidelines.
  Salvage chemotherapy included:
  Low dose cytarabine (LoDAC): 20 mg cytarabine administered twice daily by subcutaneous (SC)/intravenous (IV) injection for 10 days.
  Mitoxantrone, etoposide and intermediate dose cytarabine (MEC): mitoxantrone 6 milligrams per square meter(mg/m^2) per day administered by IV for 5 days (days 1 through 5), etoposide 100 mg/m^2 per day administered by IV for 5 days (days 1 through 5), cytarabine 1000 mg/m^2 per day administered by IV for 5 days (days 1 through 5).
  Fludarabine, cytarabine and granulocyte colony-stimulating factor (FLAG): granulocyte colony-stimulating factor (G-CSF) 300 micrograms per square meter (μg/m^2) per day administered by SC/IV for 5 days (days 1 through 5), fludarabine 30 mg/m^2 per day administered by IV for 5 days (days 2 through 6), cytarabine 2000 mg/m^2 per day administered by IV for 5 days (days 2 through 6). Participants who met treatment discontinuation criteria, entered long-term follow-up and remained in the period for up to 3 years from the participant's end of treatment visit/until discontinuation from study.
  Based on the outcome of interim analysis, at investigators discretion, participants in the treatment period had the option to enter crossover extension (COE) period to receive 120 mg gilteritinib, orally, once a day in continuous 28-day cycles until treatment discontinuation criteria was met.
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 137 | 139
Percentage of participants | 53.3 [44.6 to 61.9] | 22.3 [15.7 to 30.1]
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Treatment difference = 31.2, 95% CI 2-sided [20.2 to 42.3]

12. Secondary Outcome: Time to CRc
Description: Time to CRc (TTCRc) was defined as the time from the date of randomization until the date of first CRc.
  CRc: Rate of all complete and incomplete remissions (CR + CRp +Cri) CR: morphologically leukemia-free state, with ANC> 1x10^9/L, platelet count ≥ 100x10^9/L and normal marrow differential with <5% blasts. They were RBC and platelet transfusion independent and no evidence of extramedullary leukemia.
  CRp: met all CR criteria except incomplete platelet recovery (< 100x10^9/L). CRi: met all CR criteria, except for incomplete hematological recovery with residual neutropenia < 1x10^9/L with or without complete platelet recovery.
Time Frame: From randomization until date of first CRc (up to approximately 74 months)
Population: ITT population. Participants who achieved CRc were analyzed.
Measure: Median (Full Range); unit: months
Groups:
- Gilteritinib: Participants received 120 milligrams (mg) gilteritinib (3 tablets of 40 mg) orally, once a day in continuous 28-day cycles until treatment discontinuation criteria were met. Participants who met the treatment discontinuation criteria, entered the long-term follow-up period. Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day in continuous 28-day cycles until treatment discontinuation criteria were met. Participants who met the treatment discontinuation criteria, entered the long-term follow-up period. Participants remained in the long-term follow-up period for up to 3 years from the participant's end of treatment visit or until discontinuation from the study.
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 73 | 31
months | 1.8 [1 to 8] | 1.0 [1 to 2]

13. Secondary Outcome: Time to CR
Description: Time to CR (TTCR) was defined as the time from the date of randomization until the date of first CR.
  CR: morphologically leukemia-free state, with ANC> 1x10^9/L, platelet count ≥ 100x10^9/L and normal marrow differential with < 5% blasts. They were RBC and platelet transfusion independent and no evidence of extramedullary leukemia.
Time Frame: From randomization until date of first CR (up to approximately 74 months)
Population: ITT population. Participants who achieved CR were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 28 | 16
months | 3.7 [1 to 19] | 1.1 [1 to 2]

14. Secondary Outcome: Time to Response
Description: Time to Response (TTR) was defined as the time from the date of randomization until the date of either first response (CRc or PR).
  CRc: Rate of all complete and incomplete remissions (CR + CRp +Cri) CR: morphologically leukemia-free state, with ANC> 1x10^9/L, platelet count ≥ 100x10^9/L and normal marrow differential with <5% blasts. They were RBC and platelet transfusion independent and no evidence of extramedullary leukemia.
  CRp: met all CR criteria except incomplete platelet recovery (< 100x10^9/L). CRi: met all CR criteria, except for incomplete hematological recovery with residual neutropenia < 1x10^9/L with or without complete platelet recovery.
  PR: condition with regeneration of normal hematopoietic cells in BM, no detectable blasts, ≥ 50% decrease of blasts in BM aspirate & total BM blasts of 5-25%.
Time Frame: From randomization until date of first CRc or PR (up to approximately 74 months)
Population: ITT population. Participants who achieved CRc or PR were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 93 | 38
months | 1.0 [1 to 7] | 1.0 [1 to 2]

15. Secondary Outcome: Time to CR/CRh
Description: Time to CR/CRh (TTCRCRh) was defined as the time from the date of randomization until the date of first CR/CRh.
  CR: morphologically leukemia-free state, with ANC> 1x10^9/L, platelet count ≥ 100x10^9/L and normal marrow differential with <5% blasts. They were RBC and platelet transfusion independent and no evidence of extramedullary leukemia.
  CRh was defined as a condition at the post baseline visit, having bone marrow blasts < 5%, partial hematologic recovery ANC ≥ 0.5x10^9/L and platelets ≥ 50x10^9/L, no evidence of extramedullary leukemia and cannot be classified as CR. The blast counts in peripheral blood was ≤ 2%.
Time Frame: From randomization until date of first CR/CRh (up to approximately 74 months)
Population: ITT population. Participants who achieved CR/CRh were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 44 | 20
months | 2.8 [1 to 11] | 1.1 [1 to 2]

16. Secondary Outcome: Percentage of Participants With Transfusion Conversion and Transfusion Maintenance
Description: Transfusion conversion rate: Percentage of transfusion dependent participants at baseline period but became transfusion independent at post-baseline period divided by total participants who were transfusion dependent at baseline period.
  Transfusion maintenance rate: Percentage of transfusion independent participants at baseline period and still maintained transfusion independent at post-baseline period divided by total participants who were transfusion independent at baseline period.
  Baseline transfusion status: Participants were classified as transfusion independent if there were no RBC or platelet transfusions within 28 days prior to first dose to 28 days after first dose; otherwise classified as transfusion dependent.
  Post baseline transfusion status: Participants on treatment ≥ 84 days were classified as transfusion independent, if consecutive 56 days without any RBC or platelet transfusion; otherwise classified as transfusion dependent
Time Frame: Baseline up to approximately 74 months
Population: ITT population with available data at specified timepoint. This endpoint was planned to be analyzed only for Giltertinib arm.
Measure: Number; unit: Percentage of participants
Arm/Group | Gilteritinib
Number analyzed (Participants) | 137
Percentage of participants
  Transfusion Conversion Rate: number analyzed (Participants) | 110
  Transfusion Conversion Rate | 42.7
  Transfusion Maintenance Rate: number analyzed (Participants) | 24
  Transfusion Maintenance Rate | 70.8

17. Secondary Outcome: Percentage of Participants With Transplantation Rate
Description: Transplantation rate is defined as the percentage of participants undergoing Hematopoietic stem cell transplant (HSCT) during the study period.
Time Frame: Baseline up to approximately 74 months
Population: ITT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 137 | 139
Percentage of participants | 22.6 [15.9 to 30.6] | 7.9 [4.0 to 13.7]
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Test type: Superiority; p = 0.00055, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Treatment difference = 14.7, 95% CI 2-sided [6.5 to 22.8]

18. Secondary Outcome: Change From Baseline in Brief Fatigue Inventory (BFI)
Description: The BFI is a screening tool designed to assess the severity and impact of fatigue on daily functioning of participants with cancer during the 24 hours. There are 9 items on the scale. The first three questions ask participants to rate their fatigues on a scale from 0 (no fatigue) - 10 (as bad as you can imagine), with higher scores indicating worse outcome. The remaining six questions ask participants to rate how much fatigue has interfered with their daily activities on a scale from 0 (Does not interfere) to 10 (Completely interferes). A global fatigue score can be obtained by averaging all the items on the BFI, ranging between 0 to 10; a higher BFI fatigue score indicates worse outcome. The global BFI scores were calculated only if at least 5 of the 9 items are answered.
Time Frame: Baseline, End of treatment (63 months)
Population: ITT population with data available at specified timepoint.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 84 | 89
Scores on scale | 1.42 (2.99) | 0.75 (2.92)
Statistical Analysis 1: Comparison: Gilteritinib vs Salvage Chemotherapy; Test type: Superiority; p = 0.14841, ANCOVA — Analysis of covariance (ANCOVA) including treatment as a fixed factor, baseline score, response to first-line AML therapy and preselected salvage chemotherapy per IRT as covariates. LS Mean difference was estimated using chemotherapy as control; Least square mean difference = 0.6

19. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE could therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. TEAE was defined as an adverse event observed after starting administration of the study drug.
Time Frame: From the date of first dose up to approximately 74 months
Population: Safety Analysis Set (SAF): The SAF consisted of all participants who received at least 1 dose of study treatment (gilteritinib or salvage chemotherapy).
Measure: Number; unit: Participants
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 134 | 119
Participants | 134 | 119

20. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Scores
Description: The ECOG Scale was used to assess performance status. Number of participants with each grade was reported.
  Grade Description:
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. Dead.
Time Frame: Baseline, end of treatment visit (63 months)
Population: SAF population with available data at specified timepoint.
Measure: Number; unit: Participants
Arm/Group | Gilteritinib | Salvage Chemotherapy
Number analyzed (Participants) | 134 | 119
Participants
  Grade 0 at baseline | 35 | 37
  Grade 1 at baseline | 65 | 64
  Grade 2 at baseline | 34 | 18
  Grade 3 at baseline | 0 | 0
  Grade 4 at baseline | 0 | 0
  Grade 5 at baseline | 0 | 0
  Grade 0 at End of Treatment: number analyzed (Participants) | 83 | 94
  Grade 0 at End of Treatment | 17 | 26
  Grade 1 at End of Treatment: number analyzed (Participants) | 83 | 94
  Grade 1 at End of Treatment | 36 | 39
  Grade 2 at End of Treatment: number analyzed (Participants) | 83 | 94
  Grade 2 at End of Treatment | 19 | 21
  Grade 3 at End of Treatment: number analyzed (Participants) | 83 | 94
  Grade 3 at End of Treatment | 10 | 6
  Grade 4 at End of Treatment: number analyzed (Participants) | 83 | 94
  Grade 4 at End of Treatment | 1 | 2
  Grade 5 at End of Treatment: number analyzed (Participants) | 83 | 94
  Grade 5 at End of Treatment | 0 | 0

21. Secondary Outcome: Pharmacokinetics (PK) of Gilteritinib in Chinese PK Cohort: Area Under the Concentration Curve at 24 Hours (AUC24)
Description: AUC24 was derived from the PK samples collected.
Time Frame: Cycle 1 Day 1(C1D1): predose, 0.5, 1, 2, 3, 4, 6, 10, 24 hour post dose, Cycle 1 Day 15(C1D15): predose, 0.5, 1, 2, 3, 4, 6, 10, 24 hour post dose
Population: Pharmacokinetics Analysis Set (PKAS): The PKAS consisted of all participants who received at least 1 administration of study intervention for which at least 1 concentration data with time of dosing and sampling were available. This endpoint was planned to be analyzed only for participants in Giltertinib PK cohort which included 21 participants from six china sites.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliters(ng*h/mL)
Arm/Group | Gilteritinib
Number analyzed (Participants) | 21
nanogram*hour per milliliters(ng*h/mL)
  C1D1 | 3230 (1970)
  C1D15: number analyzed (Participants) | 16
  C1D15 | 10000 (6670)

22. Secondary Outcome: PK of Gilteritinib in Chinese PK Cohort: Maximum Concentration (Cmax)
Description: Cmax was derived from the PK samples collected.
Time Frame: C1D1: predose, 0.5, 1, 2, 3, 4, 6, 10, 24 hour post dose, C1D15: predose, 0.5, 1, 2, 3, 4, 6, 10, 24 hour post dose
Population: PKAS. This endpoint was planned to be analysed only for participants in Giltertinib PK cohort which included 21 participants from six china sites.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Gilteritinib
Number analyzed (Participants) | 21
ng/mL
  C1D1 | 206 (112)
  C1D15: number analyzed (Participants) | 16
  C1D15 | 536 (323)

23. Secondary Outcome: PK of Gilteritinib: Observed Trough Concentration (Ctrough)
Description: Ctrough was derived from the PK samples collected.
Time Frame: Predose on C1D15
Population: PKAS with available data at timepoint were analyzed. This endpoint was planned to be analyzed only for participants at the China site in the Giltertinib PK cohort.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Gilteritinib
Number analyzed (Participants) | 15
ng/mL | 323 (222)

24. Secondary Outcome: PK of Gilteritinib in Chinese PK Cohort: Time to Maximum Concentration (Tmax)
Description: tmax was derived from the PK samples collected.
Time Frame: C1D1: predose, 0.5, 1, 2, 3, 4, 6, 10, 24 hours (+/- 20 minutes) post dose, C1D15: predose, 0.5, 1, 2, 3, 4, 6, 10, 24 hours (+/- 20 minutes) post dose
Population: as for outcome 22
Measure: Median (Full Range); unit: hours
Arm/Group | Gilteritinib
Number analyzed (Participants) | 21
hours
  Cycle 1 Day 1 | 4.00 [2.00 to 24.1]
  Cycle 1 Day 15: number analyzed (Participants) | 16
  Cycle 1 Day 15 | 3.85 [1.00 to 24.3]

25. Secondary Outcome: Ctrough Concentration of Gilteritinib
Description: Concentrations below the lower limit of quantification (0.5 ng/mL) were set to zero.
Time Frame: Predose C1D8, C1D15, Day 1 of each cycle from C2 to C65, C67D1,C68D1,C69D1,C70D1
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Gilteritinib
Number analyzed (Participants) | 137
ng/mL
  C1D8: number analyzed (Participants) | 110
  C1D8 | 310 (177)
  CID15: number analyzed (Participants) | 113
  CID15 | 367 (243)
  C2D1: number analyzed (Participants) | 106
  C2D1 | 425 (305)
  C3D1: number analyzed (Participants) | 100
  C3D1 | 457 (358)
  C4D1: number analyzed (Participants) | 83
  C4D1 | 420 (428)
  C5D1: number analyzed (Participants) | 67
  C5D1 | 407 (487)
  C6D1: number analyzed (Participants) | 51
  C6D1 | 284 (275)
  C7D1: number analyzed (Participants) | 44
  C7D1 | 370 (477)
  C8D1: number analyzed (Participants) | 39
  C8D1 | 328 (323)
  C9D1: number analyzed (Participants) | 31
  C9D1 | 351 (381)
  C10D1: number analyzed (Participants) | 28
  C10D1 | 322 (383)
  C11D1: number analyzed (Participants) | 23
  C11D1 | 336 (426)
  C12D1: number analyzed (Participants) | 23
  C12D1 | 460 (703)
  C13D1: number analyzed (Participants) | 21
  C13D1 | 368 (409)
  C14D1: number analyzed (Participants) | 19
  C14D1 | 386 (449)
  C15D1: number analyzed (Participants) | 14
  C15D1 | 396 (541)
  C16D1: number analyzed (Participants) | 12
  C16D1 | 200 (116)
  C17D1: number analyzed (Participants) | 11
  C17D1 | 228 (138)
  C18D1: number analyzed (Participants) | 9
  C18D1 | 201 (143)
  C19D1: number analyzed (Participants) | 14
  C19D1 | 231 (270)
  C20D1: number analyzed (Participants) | 9
  C20D1 | 241 (190)
  C21D1: number analyzed (Participants) | 12
  C21D1 | 221 (112)
  C22D1: number analyzed (Participants) | 8
  C22D1 | 238 (149)
  C23D1: number analyzed (Participants) | 9
  C23D1 | 152 (137)
  C24D1: number analyzed (Participants) | 11
  C24D1 | 188 (141)
  C25D1: number analyzed (Participants) | 10
  C25D1 | 192 (137)
  C26D1: number analyzed (Participants) | 9
  C26D1 | 264 (138)
  C27D1: number analyzed (Participants) | 11
  C27D1 | 199 (145)
  C28D1: number analyzed (Participants) | 11
  C28D1 | 243 (141)
  C29D1: number analyzed (Participants) | 8
  C29D1 | 184 (138)
  C30D1: number analyzed (Participants) | 9
  C30D1 | 340 (472)
  C31D1: number analyzed (Participants) | 6
  C31D1 | 426 (606)
  C32D1: number analyzed (Participants) | 6
  C32D1 | 301 (395)
  C33D1: number analyzed (Participants) | 6
  C33D1 | 431 (646)
  C34D1: number analyzed (Participants) | 6
  C34D1 | 405 (590)
  C35D1: number analyzed (Participants) | 7
  C35D1 | 298 (420)
  C36D1: number analyzed (Participants) | 7
  C36D1 | 264 (343)
  C37D1: number analyzed (Participants) | 7
  C37D1 | 437 (823)
  C38D1: number analyzed (Participants) | 4
  C38D1 | 78.0 (76.3)
  C39D1: number analyzed (Participants) | 4
  C39D1 | 107 (91.3)
  C40D1: number analyzed (Participants) | 4
  C40D1 | 114 (59.2)
  C41D1: number analyzed (Participants) | 6
  C41D1 | 152 (123)
  C42D1: number analyzed (Participants) | 8
  C42D1 | 128 (150)
  C43D1: number analyzed (Participants) | 8
  C43D1 | 96.9 (114)
  C44D1: number analyzed (Participants) | 4
  C44D1 | 148 (145)
  C45D1: number analyzed (Participants) | 4
  C45D1 | 166 (97.9)
  C46D1: number analyzed (Participants) | 5
  C46D1 | 105 (127)
  C47D1: number analyzed (Participants) | 5
  C47D1 | 116 (104)
  C48D1: number analyzed (Participants) | 5
  C48D1 | 131 (107)
  C49D1: number analyzed (Participants) | 5
  C49D1 | 74.4 (82.0)
  C50D1: number analyzed (Participants) | 5
  C50D1 | 134 (119)
  C51D1: number analyzed (Participants) | 4
  C51D1 | 130 (136)
  C52D1: number analyzed (Participants) | 3
  C52D1 | 93.4 (114)
  C53D1: number analyzed (Participants) | 3
  C53D1 | 148 (188)
  C54D1: number analyzed (Participants) | 3
  C54D1 | 166 (246)
  C55D1: number analyzed (Participants) | 3
  C55D1 | 129 (169)
  C56D1: number analyzed (Participants) | 3
  C56D1 | 157 (227)
  C57D1: number analyzed (Participants) | 1
  C57D1 | 380
  C58D1: number analyzed (Participants) | 1
  C58D1 | 338
  C59D1: number analyzed (Participants) | 1
  C59D1 | 451
  C60D1: number analyzed (Participants) | 1
  C60D1 | 362
  C61D1: number analyzed (Participants) | 1
  C61D1 | 292
  C62D1: number analyzed (Participants) | 1
  C62D1 | 287
  C63D1: number analyzed (Participants) | 1
  C63D1 | 411
  C64D1: number analyzed (Participants) | 0
  C65D1: number analyzed (Participants) | 1
  C65D1 | 362
  C67D1: number analyzed (Participants) | 1
  C67D1 | 326
  C68D1: number analyzed (Participants) | 1
  C68D1 | 584
  C69D1: number analyzed (Participants) | 1
  C69D1 | 345
  C70D1: number analyzed (Participants) | 1
  C70D1 | 313

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization up to 74 months AEs: From first dose up to 74 months
Description: All- cause mortality: ITT consisted of all participants who were randomized.
  AEs: SAF consisted of all participants who received at least 1 dose of study treatment (gilteritinib or salvage chemotherapy).
Arm/Group | Gilteritinib | Salvage Chemotherapy
All-Cause Mortality (participants affected / at risk) | 97/137 | 85/139
Serious Adverse Events (participants affected / at risk) | 102/134 | 71/119
Other Adverse Events (participants affected / at risk) | 133/134 | 113/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilteritinib (N=134) | Salvage Chemotherapy (N=119)
Agranulocytosis (Blood and lymphatic system disorders) | 4 (14) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 14 (19) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 29 (50) | 25 (30)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (35) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (4) | 4 (4)
Cardiac failure (Cardiac disorders) | 2 (5) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (5) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (4)
Small intestine ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 12 (13) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute graft versus host disease (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1)
Chronic graft versus host disease in liver (Immune system disorders) | 1 (1) | 0 (0)
Graft versus host disease in eye (Immune system disorders) | 1 (1) | 0 (0)
Acinetobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Candida sepsis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 3 (4) | 1 (1)
Fungal infection (Infections and infestations) | 2 (3) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (4) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 2 (2) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic infection (Infections and infestations) | 2 (2) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 8 (16) | 4 (5)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Oral infection (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngeal abscess (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 24 (41) | 8 (10)
Pseudomonal sepsis (Infections and infestations) | 1 (2) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 9 (14) | 15 (17)
Septic shock (Infections and infestations) | 5 (9) | 5 (8)
Skin infection (Infections and infestations) | 7 (8) | 0 (0)
Soft tissue infection (Infections and infestations) | 2 (2) | 1 (1)
Toxic shock syndrome (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (10)
Platelet count decreased (Investigations) | 3 (7) | 1 (5)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 1 (1) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 1 (2) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 2 (4)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (2) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (3)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (3) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilteritinib (N=134) | Salvage Chemotherapy (N=119)
Anaemia (Blood and lymphatic system disorders) | 99 (719) | 79 (394)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4) | 8 (11)
Leukocytosis (Blood and lymphatic system disorders) | 25 (53) | 14 (18)
Leukopenia (Blood and lymphatic system disorders) | 41 (465) | 32 (199)
Lymphopenia (Blood and lymphatic system disorders) | 11 (77) | 14 (103)
Neutropenia (Blood and lymphatic system disorders) | 41 (414) | 24 (95)
Thrombocytopenia (Blood and lymphatic system disorders) | 56 (594) | 44 (314)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 9 (10)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 7 (7)
Constipation (Gastrointestinal disorders) | 19 (29) | 15 (19)
Diarrhoea (Gastrointestinal disorders) | 40 (61) | 28 (41)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 (7) | 2 (3)
Gingival bleeding (Gastrointestinal disorders) | 7 (7) | 5 (6)
Mouth haemorrhage (Gastrointestinal disorders) | 7 (14) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 18 (23) | 9 (10)
Nausea (Gastrointestinal disorders) | 24 (33) | 31 (42)
Vomiting (Gastrointestinal disorders) | 25 (33) | 30 (43)
Asthenia (General disorders) | 13 (14) | 10 (12)
Fatigue (General disorders) | 7 (7) | 6 (7)
Oedema peripheral (General disorders) | 12 (13) | 3 (4)
Pyrexia (General disorders) | 54 (149) | 45 (96)
Hepatic function abnormal (Hepatobiliary disorders) | 13 (36) | 3 (6)
Febrile infection (Infections and infestations) | 7 (10) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 9 (10) | 5 (5)
Oral infection (Infections and infestations) | 2 (7) | 7 (9)
Pneumonia (Infections and infestations) | 34 (46) | 23 (27)
Skin infection (Infections and infestations) | 9 (10) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 26 (47) | 8 (8)
Urinary tract infection (Infections and infestations) | 7 (7) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 7 (7) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 7 (8) | 2 (2)
Alanine aminotransferase increased (Investigations) | 49 (200) | 23 (41)
Aldolase increased (Investigations) | 8 (10) | 0 (0)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 11 (17) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 56 (182) | 19 (32)
Blood albumin decreased (Investigations) | 7 (8) | 5 (11)
Blood alkaline phosphatase increased (Investigations) | 26 (74) | 7 (17)
Blood bilirubin increased (Investigations) | 21 (54) | 14 (30)
Blood creatine phosphokinase MB increased (Investigations) | 10 (26) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 36 (82) | 1 (4)
Blood creatinine increased (Investigations) | 13 (22) | 2 (4)
Blood fibrinogen decreased (Investigations) | 11 (18) | 5 (8)
Blood lactate dehydrogenase increased (Investigations) | 61 (139) | 22 (38)
C-reactive protein increased (Investigations) | 20 (147) | 11 (54)
Electrocardiogram QT prolonged (Investigations) | 12 (18) | 0 (0)
Eosinophil count decreased (Investigations) | 3 (10) | 10 (17)
Eosinophil percentage decreased (Investigations) | 5 (41) | 9 (34)
Fibrin D dimer increased (Investigations) | 14 (38) | 4 (6)
Gamma-glutamyltransferase increased (Investigations) | 27 (108) | 9 (23)
Lymphocyte count decreased (Investigations) | 28 (260) | 27 (162)
Lymphocyte count increased (Investigations) | 7 (21) | 9 (16)
Lymphocyte percentage decreased (Investigations) | 7 (29) | 17 (49)
Lymphocyte percentage increased (Investigations) | 10 (43) | 19 (38)
Monocyte count decreased (Investigations) | 10 (51) | 16 (38)
Monocyte count increased (Investigations) | 7 (23) | 13 (24)
Monocyte percentage decreased (Investigations) | 7 (19) | 13 (36)
Monocyte percentage increased (Investigations) | 6 (31) | 19 (35)
Neutrophil count decreased (Investigations) | 51 (579) | 44 (239)
Neutrophil count increased (Investigations) | 11 (14) | 8 (9)
Neutrophil percentage decreased (Investigations) | 10 (51) | 21 (61)
Neutrophil percentage increased (Investigations) | 3 (17) | 8 (12)
Platelet count decreased (Investigations) | 55 (858) | 50 (462)
Procalcitonin increased (Investigations) | 10 (25) | 1 (1)
Weight decreased (Investigations) | 12 (18) | 11 (12)
Weight increased (Investigations) | 33 (68) | 1 (1)
White blood cell count decreased (Investigations) | 55 (604) | 51 (250)
White blood cell count increased (Investigations) | 9 (14) | 13 (17)
Decreased appetite (Metabolism and nutrition disorders) | 8 (10) | 7 (9)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 (19) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 36 (82) | 18 (39)
Hypermagnesaemia (Metabolism and nutrition disorders) | 7 (18) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 17 (66) | 7 (13)
Hyperuricaemia (Metabolism and nutrition disorders) | 12 (30) | 11 (11)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 26 (89) | 23 (48)
Hypocalcaemia (Metabolism and nutrition disorders) | 37 (130) | 26 (70)
Hypokalaemia (Metabolism and nutrition disorders) | 57 (140) | 45 (117)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (14) | 13 (21)
Hyponatraemia (Metabolism and nutrition disorders) | 29 (93) | 23 (57)
Hypophosphataemia (Metabolism and nutrition disorders) | 20 (34) | 7 (24)
Hypoproteinaemia (Metabolism and nutrition disorders) | 24 (107) | 10 (30)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (16) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (11) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (1)
Dizziness (Nervous system disorders) | 14 (19) | 5 (6)
Headache (Nervous system disorders) | 12 (13) | 6 (6)
Insomnia (Psychiatric disorders) | 12 (14) | 6 (6)
Haematuria (Renal and urinary disorders) | 11 (12) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 9 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 (30) | 8 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (14) | 6 (6)
Petechiae (Skin and subcutaneous tissue disorders) | 7 (14) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 21 (39) | 12 (13)
Hypertension (Vascular disorders) | 24 (72) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT03182244/Prot_002.pdf
  • Statistical Analysis Plan (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT03182244/SAP_003.pdf